CLINICAL TRIAL: NCT00637754
Title: Safety of Sports for Patients With Implantable Cardioverter-Defibrillators: A Multi-Center Registry
Brief Title: Safety of Sports for Patients With Implantable Cardioverter-Defibrillators
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Medtronic (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Rachel Lampert, Principal Investigator, Yale University
Other Study IDs: 0608001730
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Heart Arrhythmias
Keywords: ICD; Sports
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The registry will obtain information to determine the safety of sports participation for patients with defibrillators (ICDs).

DETAILED DESCRIPTION:
Patients who are participating in sports who have defibrillators will be invited to participate in a prospective registry to determine the rate of adverse events occurring during sporting activities. Patients will be followed for four years and adverse events quantified. Yale is the coordinating center for this multicenter registry.

ELIGIBILITY:
Inclusion Criteria:

* individuals between the ages of 10 and 60
* has a defibrillator
* plays a competitive/organized sport more vigorous than golf or bowling or participates in a dangerous sport

Exclusion Criteria:

* children under 10 years (as they engage in primarily recreational sports)
* individuals over the age of 60 years (maintain a homogenous population)
* inability to give informed consent

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals between the ages of 10 and 60 years who have defibrillators who participate in competitive (organized sports at any level) or dangerous sports.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2006-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Resuscitated arrest or death during sports, or injury during sports due to arrhythmic symptoms and/or shock. | four years

SECONDARY OUTCOMES:
System malfunction and incidence of ventricular arrhythmias (VA) requiring multiple shocks for termination | four years.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lampert, MD, Principal Investigator — Yale University
Locations (54):
- United States (31):
  - Arizona Pediatric Cardiology Consultants, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Foundation for the Advancement of Cardiovascular Therapy, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Arrhythmia Center of Connecticut, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Cypress Heart, Wichita, Kansas
  - Midatlantic Cardiovascular Associates, PA, Towson, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Michigan Heart, PC, Ann Arbor, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Park Nicollet, Minneapolis, Minnesota
  - Children's Hospital and Clinics of Minnesota, Roseville, Minnesota
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Research Foundation, Columbus, Ohio
  - Legacy Cllinical Research & Tech Center (Good Samaritan Hospital_, Portland, Oregon
  - Main Line Health Heart Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- St. Vincent's Hospital, Mebourne LTD, Fitzroy, Victoria, Australia
- Belgium (4):
  - OLV Hospital Aalst, Aalst
  - Clin.du sud-Luxembourg, Arlon
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
- Canada (3):
  - The University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre University Hospital, London, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
- IKEM, Prague, Czechia
- France (2):
  - CHRU-Hopital de Pontchaillou, Rennes
  - Dlinique Pasteur, Toulouse
- Germany (2):
  - Univeristy of Leipzig Heart Centre, Leipzig
  - Klinikum Bogenhausen, München
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Netherlands (2):
  - Radboud University Hospital Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Rikshospitalet Oslo, Oslo, Norway
- Sterling Memorial University Hospital, Lodz, Poland
- Spain (2):
  - Hospital Clinic-University of Barcelona, Barcelona
  - Hospital Puerta de Hierro, Majadahonda
- Switzerland (2):
  - University of Bern, Bern
  - University Hospital Zurich, Zurich
- Southampton General Hospital, Hants, United Kingdom

REFERENCES:
- [Derived] Saarel EV, Law I, Berul CI, Ackerman MJ, Kanter RJ, Sanatani S, Cohen MI, Berger S, Fischbach PS, Burton DA, Dziura J, Brandt C, Simone L, Li F, Olshansky B, Cannom DS, Lampert RJ. Safety of Sports for Young Patients With Implantable Cardioverter-Defibrillators: Long-Term Results of the Multinational ICD Sports Registry. Circ Arrhythm Electrophysiol. 2018 Nov;11(11):e006305. doi: 10.1161/CIRCEP.118.006305. PMID 30520349